CLINICAL TRIAL: NCT02564081
Title: Remote Effects of Lower Limb Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SpM2015-001
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Fascia; Randomized Controlled Trial; Stretching; Myofascial

ARMS (3):
- Static Stretching lower limb (Experimental): Three 30 s bouts of static stretching for the gastrocnemius and the hamstrings respectively
  Interventions: Other: Static Stretching lower limb
- Static stretching Cervical (Active Comparator): Six 30 s bouts of static stretching of the cervical spine in the sagittal plane (flexion only)
  Interventions: Other: Static stretching Cervical
- Ctrl (No Intervention): No intervention

INTERVENTIONS:
Other: Static Stretching lower limb
  Arms: Static Stretching lower limb
Other: Static stretching Cervical
  Arms: Static stretching Cervical

SUMMARY:
Recent research suggests that the skeletal muscles and the fibrous connective tissue form a body-wide network of myofascial chains. A systematic analysis of dissection studies suggests that fascia links at least a variety of muscles to myofascial chains (Wilke et al. 2015). As fascia can modify its stiffness, strain transmission along these meridians is supposable (Norton-Old et al. 2013). Tensile transmission along myofascial chains might contribute to the proper functioning of the movement system. However, despite solid evidence from in vitro studies, scarce data is available concerning the in vivo behavior of the meridians. The present study is conducted to resolve this research deficit and to elucidate whether stretching of the lower limb muscles increases neck mobility. Healthy subjects (n = 3 x 20) participate in the randomized controlled trial. One group performs three 30 s bouts of static stretching for the gastrocnemius and the hamstrings respectively. A control group remains inactive for the same time. Participants of the third group perform 6x30 s bouts of static stretching of the cervical spine in zhe sagittal plane (flexion only). Pre and post intervention as well as 5 min after the intervention, maximal cervical range of motion (ROM) in flexion/extension, lateral flexion and rotation was assessed using an ultrasonic movement analysis system.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants after subscribing informed consent

Exclusion Criteria:

* severe orthopedic, cardiovascular, neurological, psychiatric or endocrine diseases, not completely healed traumata, drug intake in the past 48 hours, pregnancy and presence of muscle soreness.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximal cervical range of motion in flexion/extension | 2 min.

SECONDARY OUTCOMES:
Maximal cervical range of motion in lateral flexion | 2 min.
Maximal cervical range of motion in rotation | 2 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Goethe University Frankfurt/Main, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Wilke J, Krause F, Vogt L, Banzer W. What Is Evidence-Based About Myofascial Chains: A Systematic Review. Arch Phys Med Rehabil. 2016 Mar;97(3):454-61. doi: 10.1016/j.apmr.2015.07.023. Epub 2015 Aug 14. PMID 26281953
- [Background] Norton-Old KJ, Schache AG, Barker PJ, Clark RA, Harrison SM, Briggs CA. Anatomical and mechanical relationship between the proximal attachment of adductor longus and the distal rectus sheath. Clin Anat. 2013 May;26(4):522-30. doi: 10.1002/ca.22116. Epub 2012 Jun 14. PMID 23553712